CLINICAL TRIAL: NCT03614845
Title: Evaluation of Effect of Different Ventilator Mods on Atelectasis in Patients Undergoing Laparoscopic Surgery: a Prospective Randomized Controlled Clinical Trial
Brief Title: Evaluation of Effect of Different Ventilator Mods on Atelectasis in Patients Undergoing Laparoscopic Surgery
Acronym: PCV-VG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse Zeynep Turan, Principal Investigator, Derince Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DerinceTRH-006
Record Dates: First submitted 2018-07-22; First posted 2018-08-03 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Atelectasis; Atelectases, Postoperative Pulmonary
Keywords: postoperative atelectasis; mechanical ventilation; laparoscopic surgery; lung ultrasonography; volume controlled ventilation; pressure controlled
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VCV-Lung Ultrasonography (Active Comparator): patients undergoing laparoscopic surgery will be performed pre and postoperatively lung ultrasonography. after induction of anesthesia patients will be supported by mechanical ventilation on volume controlled ventilation mode.
  Interventions: Procedure: VCV; Diagnostic Test: lung ultrasonography
- PCV-VG- Lung Ultrasonography (Active Comparator): patients undergoing laparoscopic surgery will be performed pre and postoperatively lung ultrasonography.after induction of anesthesia patients will be supported by mechanical ventilation on pressure controlled volume guaranteed mode
  Interventions: Procedure: PCV-VG; Diagnostic Test: lung ultrasonography

INTERVENTIONS:
Procedure: VCV — after induction for anesthesia patients will be supported by mechanical ventilation on volume controlled ventilation mode
  Arms: VCV-Lung Ultrasonography
Procedure: PCV-VG — after induction for anesthesia patients will be supported by mechanical ventilation on pressure controlled and volume guaranteed ventilation mode
  Arms: PCV-VG- Lung Ultrasonography
Diagnostic Test: lung ultrasonography — all patients will be performed lung ultrasonography pre and postoperatively

SUMMARY:
In this study researchers aim to evaluate effect of different ventilation modalities on the developments of atelectasis by using ultrasound.

DETAILED DESCRIPTION:
Patients undergoing laparoscopic surgery will be randomly assigned either volume controlled ventilation group or pressure controlled volume guaranteed ventilation group. All patients will be performed lung ultrasonography pre and postoperatively to evaluate the development of lung atelectasis and effect of different ventilation modalities on the development of atelectasis.

ELIGIBILITY:
Inclusion Criteria:

* undergoing laparoscopic surgery
* ASA Status I-II

Exclusion Criteria:

* Gastroesophageal reflux
* obstructive sleep apnea syndrome
* BMI>30
* severe lung and heart disease
* ASA Status III-IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Effect of different ventilation mods on development of peroperative atelectasis | at minute 5 in postoperative care unit
  Patients undergoing laparoscopic surgery will be assigned either volume controlled mode or pressure support volume guaranteed mode. After the operation a researcher will perform lung ultrasonography postoperative at minute 5. Researcher will detect 6 region of each lung totally 12 regions . The researcher will record the modified and original lung ultrasonography scores (LUS Score) of the patients. LUS Score is a scoring system to evaluate atelectasis of lung and scores 1-3 points for each region (Min score 0 max score 36)

SECONDARY OUTCOMES:
Effect of different ventilation mods on development of peroperative atelectasis | at minute 30 in postoperative care unit
  Patients undergoing laparoscopic surgery will be assigned either volume controlled mode or pressure support volume guaranteed mode. After the operation a researcher will perform lung ultrasonography in postoperative care unit at minute 30. Researcher will detect 6 region of each lung totally 12 regions . The researcher will record the modified and original lung ultrasonography scores (LUS Score) of the patients. LUS Score is a scoring system to evaluate atelectasis of lung and scores 1-3 points for each region.(Min score 0 max score 36)

CONTACTS AND LOCATIONS:
Overall Officials: Ayten Saracoglu, Study Director — Marmara Unıversity Medical Sciences
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University School of Medicine, Istanbul
  - Derince Research and Training Hospital, Kocaeli